CLINICAL TRIAL: NCT04522336
Title: A Pilot Trial of Pembrolizumab Plus Chemoradiotherapy in Participants With Unresectable Gastroesophageal Cancer
Brief Title: Pembrolizumab and Chemoradiotherapy for the Treatment of Unresectable Gastroesophageal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1253; NCI-2020-05251 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1253 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-03

CONDITIONS: Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Localized Gastroesophageal Junction Adenocarcinoma; Locally Advanced Gastroesophageal Junction Adenocarcinoma; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Unresectable Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Docetaxel; Fluorouracil; dehydroftorafur; Oxaliplatin; pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, chemoradiotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Docetaxel; Drug: Fluorouracil; Drug: Oxaliplatin; Biological: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Receive radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial investigates how well pembrolizumab and chemoradiotherapy works in treating patients with gastroesophageal cancer that cannot be removed by surgery (unresectable). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as fluorouracil, oxaliplatin and docetaxel work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy photons to kill tumor cells and shrink tumors. Giving pembrolizumab together with chemoradiotherapy may help to control gastroesophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the clinical activity (as assessed by complete clinical response rate) of pembrolizumab plus chemoradiation.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of pembrolizumab plus chemoradiation.

II. To determine the overall survival efficacy of pembrolizumab plus chemoradiation.

III. Evaluate progression free survival (PFS) by local investigator review and by blinded central radiologists' review.

EXPLORATORY OBJECTIVES:

I. To explore the association between PD-L1 expression by immunohistochemistry, somatic gene expression profiling, and clinical efficacy of pembrolizumab.

II. To explore the relationship between genomic variation and response to study treatment.

III. To identify molecular (genomic, metabolic, and/or proteomic) biomarkers that may correlate with clinical response/resistance, safety, pharmacodynamic activity, and/or the mechanism of action of pembrolizumab in combination with chemoradiation.

IV. To determine the effect of pembrolizumab plus chemoradiation treatment on tumor T cell infiltration.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment with pembrolizumab repeats every 3 weeks for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive oxaliplatin IV over 2 hours on day 1 followed by fluorouracil IV over 48 hours once every 2 weeks (Q2W) for 8 weeks (4 cycles) in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION CHEMORADIATION: After a 3 week treatment free period, patients receive pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive fluorouracil IV continuous over 5 days (Monday through Friday) for 5 weeks and docetaxel IV over 1 hour once a week (QW) for 5 weeks in the absence of disease progression or unacceptable toxicity. Starting no later than 3 days after the beginning of the Consolidation Chemoradiation period, patients also undergo 28 fractions of radiation therapy in the absence of disease progression or unacceptable toxicity.

After a 6-9 week treatment free period, patients continue pembrolizumab IV over 30 minutes on day 1. Treatment with pembrolizumab repeats every 3 weeks for up to 30 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 9-12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed diagnosis of unresectable gastroesophageal adenocarcinoma will be enrolled in this study for systemic treatment first
* Have histologically documented locally advanced unresectable cancer or localized cancer in a patient who declines surgery
* Participant is able to provide endoscopic research biopsies and research blood
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 7 days prior to treatment initiation
* A male participant must agree to use a contraception during the treatment period and for at least 120 days, corresponding to time needed to eliminate any study treatment(s) after the last dose of study treatment and refrain from donating sperm during this period
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days/weeks after the last dose of study treatment
* Patients with stable brain metastasis and/or carcinomatous leptomeningeal disease as defined in exclusion criteria
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial. The participant may also provide consent for future biomedical research. However, the participant may participate in the main trial without participating in future biomedical research
* Absolute neutrophil count >= 1500/uL (within 10 days prior to the start of study treatment)
* Platelets >= 100 000/uL (within 10 days prior to the start of study treatment)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (within 10 days prior to the start of study treatment)

  * Criteria may be met with blood transfusion as these tumors are losing blood
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated* creatinine clearance (CrCl) >= 60 mL/min for participant with creatinine levels > 1.5 x institutional ULN (within 10 days prior to the start of study treatment) (GFR can also be used in place of creatinine or CrCl)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =<1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN (within 10 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (within 10 days prior to the start of study treatment)
* International normalized ratio (INR) OR prothrombin time (PT), activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 10 days prior to the start of study treatment)

Exclusion Criteria:

* Has cancer that is confined to the stomach and not involving gastroesophageal junction
* Has significant cardiovascular impairment within 6 months of the first dose of study drug (New York Heart Association [NYHA] class III or IV)
* Has had major surgery, open biopsy, or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of study treatment

  * Note: If participant has had major surgery, they must have recovered adequately from the toxicity and/or complications from the treatment prior to starting study intervention
* Has pre-existing peripheral neuropathy > grade 1
* Participant has a history of (non-infectious) pneumonitis that required treatment with steroids or currently has pneumonitis
* Participant has a known additional malignancy that is progressing or has required active treatment in the last 2 years

  * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, ductal carcinoma in situ, or cervical carcinoma in situ that has undergone potentially curative therapy are not excluded
* Participant has known active central nervous system (CNS) metastases and/or carcinomatous meningitis

  * Note: Participants with previously treated brain metastases may participate provided they are radiologically stable (i.e., without evidence of progression for at least 4 weeks by repeat imaging [repeat imaging should be performed during study screening]), clinically stable, and without requirement for steroid treatment for at least 14 days prior to the first dose of study treatment
* Participant has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)

  * Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment
* Participant has an active infection requiring systemic therapy
* Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's involvement for the full duration of the trial, or is not in the best interest of the participant to be involved, in the opinion of the treating investigator

  * Note: Participants who received colony-stimulating factors (e.g., granulocyte colony stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF] or recombinant erythropoietin) within 2 weeks prior to the first dose of study treatment are not eligible
* Participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Participant has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
* Participant has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection. No testing for hepatitis B or hepatitis C is required
* Participant has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T cell receptor (e.g., CTLA-4, OX 40, CD137)
* Participant has received prior systemic anti-cancer therapy including investigational agents
* Has received prior radiotherapy for the current disease
* Participant has received a live vaccine within 30 days prior to the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* Participant has severe hypersensitivity (>= grade 3) to pembrolizumab or any of its excipients
* Participant is currently participating in or has participated in a study of an investigational agent (anti-cancer agent only) or has used an investigational device within 4 weeks prior to the first dose of study treatment

  * Note: Participants who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Participant is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Participant has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis) is eligible
* Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2027-07-18 (Estimated); Study Completion 2027-07-18 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (cCR) | Up to 2 years
  cCR, defined as at the time of post-chemoradiation staging, there is no evidence of cancer on endoscopic examination/histology/cytology and there is no evidence of cancer by imaging modality. Tumor assessment will be conducted every 9 weeks until the 54th week of the study and every 12 weeks after that. The best response will be recorded.

SECONDARY OUTCOMES:
Number of participants experiencing adverse events (AEs) | Up to 90 days post treatment
  Safety and tolerability will be assessed by clinical review of all relevant parameters including AEs, laboratory tests, and vital signs. Counts and percentages of subjects with AEs will be provided.
Number of participants discontinuing study drug due to AEs | Up to 90 days post treatment
  Safety and tolerability will be assessed by clinical review of all relevant parameters including AEs, laboratory tests, and vital signs. Counts and percentages of subjects with AEs will be provided.
Overall survival (OS) | From start of treatment to death due to any cause, assessed up to 2 years
  OS will be estimated using Kaplan-Meier method.
Median progression free survival (PFS) | From date of first dose with study drug to the earliest date of progression or death by any cause (in the absence of progression), assessed up to 2 years
  PFS will be estimated using Kaplan-Meier method.
PFS at 6 months | From date of first dose with study drug to the earliest date of progression or death by any cause (in the absence of progression), assessed at 6 months
  PFS will be estimated using Kaplan-Meier method.
PFS at 12 months | From date of first dose with study drug to the earliest date of progression or death by any cause (in the absence of progression), assessed at 12 months
  PFS will be estimated using Kaplan-Meier method.
PFS at 24 months | From date of first dose with study drug to the earliest date of progression or death by any cause (in the absence of progression), assessed at 24 months
  PFS will be estimated using Kaplan-Meier method.

OTHER OUTCOMES:
Tumor PD-L1 proportion | Up to 2 years
Tumor gene expression | Up to 2 years
Tumor genetics | Up to 2 years
Biomarker analysis | Up to 2 years
Tumor T cell infiltrate | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A Ajani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT04522336/ICF_001.pdf